CLINICAL TRIAL: NCT05964179
Title: Identification of Chrononutrition Factors Associated With Chronic Non-communicable Diseases and Investigation of Circadian Gene-Chrononutrition Interactions in the Development of Chronic Non-communicable Diseases Among Koreans
Brief Title: Effects of Daily Eating Duration on Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Sangah Shin, Associated Professor, Chung-Ang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1041078-20230217-BR-035
Record Dates: First submitted 2023-07-12; First posted 2023-07-27 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Body Weight Maintenance; Nutritional and Metabolic Diseases
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- time restricted feeding (Experimental): total feeding time (from the first meal or snack to the last) is assigned as 8 hours/day.
  Interventions: Behavioral: time extended feeding
- time extended feeding (Experimental): total feeding time (from the first meal or snack to the last) is assigned as 14 hours/day.
  Interventions: Behavioral: time restricted feeding

INTERVENTIONS:
Behavioral: time extended feeding — Total feeding time (from the first meal or snack to the last meal or snack) is assigned as 14 hours per day.
  Arms: time restricted feeding
Behavioral: time restricted feeding — Total feeding time (from the first meal or snack to the last meal or snack) is assigned as 8 hours per day.
  Arms: time extended feeding

SUMMARY:
This study would recruit about 50 healthy adult women and randomly divide the participants into two groups for a ten-week crossover intervention study. The investigators aimed to observe the impact of daily feeding/fasting time on clinical metabolic biomarkers.

DETAILED DESCRIPTION:
Many nutritional epidemiological studies conducted among various population groups (Cohort study, RCT study) found that chrono-nutrition factors such as morning fasting, functional supplements like fish oils, intermittent fasting, and time-restricted feeding were related to weight management, cardiovascular metabolism, blood glucose, and blood lipid metabolism. Some dietary intervention studies have found its effect on weight loss, sleep improvement, blood glucose improvement, insulin sensitivity, β cell reactivity, blood pressure, oxidative stress, and appetite improvement. This intervention study aims to investigate changes in chronic disease risk factors according to the daily meal exposure time (from the first meal to the last meal or snack) in healthy adult women.

The subjects of this study are healthy adult women aged the 30s - 40s with a body mass index (BMI) of 23 kg/m2 or a body fat rate of 28% or higher and would be excluded if the participants have inconsistent eating patterns or weight changes of 5% or more over the past three months, are pregnant or breastfeeding, are heavy drinkers (alcohol intake of 10 g/day, 300 cc), and are smokers.

A total of 10 weeks of intervention are conducted. Two meal exposure time groups are performed for four weeks each, and there is a two-week wash-out between different exposure times. The total meal period per day would be limited to 8 hours ± 30 minutes for the TRF group, and 14 hours ± 30 minutes for the EXF group. Each group will be divided into early type (before 10 a.m.) and late type (after 10 a.m.) depending on the participants' first meal timing and will be changed to another group in the second intervention period. During the 10-week study, blood (to collect genetic information related to blood lipids, blood sugar, 10ml) and urine (to collect metabolic indicators such as urine sodium, 15ml) samples would be collected four times.

Changes in evaluation variables (body composition indicators, urine indicators, or blood indicators) before and after each intervention period will be tested using the paired t-test. The association between meal time and changes in biomarkers will be tested by ANOVA using a mixed model. The analysis would be adjusted for covariates related to lifestyle (sleeping time, physical activity level, smoking status) and chrono-nutrition-related genetic information.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult women with a body mass index (BMI) of 23 kg/m2 or a body fat rate of 28% or higher

Exclusion Criteria:

* whose eating patterns have not been consistent over the past three months who has changed his or her weight in the past three months by more than 5% who has been diagnosed with cardiovascular disease/cancer/diabetes/hypertension or who has taken drugs for related diseases be pregnant or breast-feeding within the last three months who drink too much (alcohol intake ≥ 10 g/day, about 300cc of beer, about 1 glass of soju) who smoke

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
change of body weight in kilogram before and after the intervention | before and after the two intervention periods (first intervention (baseline, week 4), second intervention ( week 7, week 10))
  Direct measurement
change of body fat in kilogram before and after the intervention | before and after the two intervention periods (first intervention (baseline, week 4), second intervention ( week 7, week 10))
  Direct measurement
change of waist circumference in centimeter before and after the intervention | before and after the two intervention periods (first intervention (baseline, week 4), second intervention ( week 7, week 10))
  Direct measurement

SECONDARY OUTCOMES:
change of fasting blood glucose (mg/dL) | before and after the two intervention periods (first intervention (baseline, week 4), second intervention ( week 7, week 10))
  Direct measurement
change of serum TG (mg/dL) | before and after the two intervention periods (first intervention (baseline, week 4), second intervention ( week 7, week 10))
  Direct measurement
change of serum HDL-C (mg/dL) | before and after the two intervention periods (first intervention (baseline, week 4), second intervention ( week 7, week 10))
  Direct measurement
change of serum TC(mg/dL) | before and after the two intervention periods (first intervention (baseline, week 4), second intervention ( week 7, week 10))
  Direct measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sangah Shin, Ph.D, Principal Investigator — Chung-Ang University
Locations (1):
- Chuang-Ang University, Anseong, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Tan LJ, Shin S. Impact of eating duration on weight management, sleeping quality, and psychological stress: A pilot study. J Nutr Biochem. 2025 Mar;137:109835. doi: 10.1016/j.jnutbio.2024.109835. Epub 2024 Dec 17. PMID 39701471